CLINICAL TRIAL: NCT01401842
Title: Reduction of Risk for Low Back Injury in Theater of Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, William Quillen, Associate Dean & Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10193004
Record Dates: First submitted 2011-06-15; First posted 2011-07-25 (Estimated); Results first posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Lower Back Injury
Keywords: low back muscular strength and endurance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strengthening Exercise (Experimental): Lumbar ext. high intensity progressive resistance exercise
  Interventions: Other: Lumbar ext. high intensity progressive resistance exercise
- Stabilization Exercise (Active Comparator): Low intensity core stabilization exercise
  Interventions: Other: Low intensity core stabilization exercise

INTERVENTIONS:
Other: Lumbar ext. high intensity progressive resistance exercise — 1 active set of 1 exercise, 1x/week, 11 weeks
  Arms: Strengthening Exercise
Other: Low intensity core stabilization exercise — 1 set of 5 exercises, 1x/week, 11 weeks
  Arms: Stabilization Exercise

SUMMARY:
The investigators will conduct a controlled clinical trial with U.S. Army soldiers training to become combat medics. The purpose of this study is to determine if a 11-week, high intensity exercise program targeting the low back muscles using specialized equipment will result in a 25% increase in low back muscular strength and endurance compared with a lower intensity general core stability exercise.

DETAILED DESCRIPTION:
Background Low back injury is responsible for the largest percentage of non-battle injuries in the theater of operations and is a large contributor to non-expiration of active service attrition in the US Armed Forces. Weakness and poor endurance of the back muscles are associated with low back injury. Targeted, high intensity exercise approaches using specialized equipment to develop the strength and endurance of the "weak link" muscle group (the lumbar extensors) have been shown to reduce risk for low back injury in high-risk civilian workers, but have not been widely implemented in military settings.

Objective/Hypothesis Specific Aim: In a controlled clinical trial, the investigators will assess the effectiveness of a high intensity progressive resistance exercise training program targeting the lumbar extensors to improve lumbar extensor muscular strength and endurance in US Army soldiers.

Hypothesis: A high intensity progressive resistance exercise for the lumbar extensors will result in a 25% increase in lumbar extensor muscular strength and endurance compared with control following the 11-week intervention.

Study Design A mixed methods, two-arm, controlled clinical trial with cluster randomization will be conducted. The sampling frame will be soldiers training to become combat medics from one domestic US Army base. Soldiers will be randomly assigned (by platoon) to one of two interventions - experimental or control. All participants at a given platoon will receive the same intervention and all interventions will be carried out at the US Army base, in addition to the soldiers' usual physical fitness training program. Participants randomized to the experimental group (strengthening exercise) will perform lumbar extensor muscle progressive resistance exercise using standardized protocols. Exercise training will consist of 1 set of high intensity progressive resistance exercise for lumbar extensors on specialized equipment. Participants in the active comparator control group (stabilization exercise) will perform 5 minutes of low intensity core stabilization exercises on the floor. Interventions will be carried out 1X/week for 11 weeks. Outcome measures that will be utilized to test the hypothesis of Aim 1 include validated physical fitness tests for lumbar extension muscular strength and endurance. Fitness tests will be conducted at baseline and following the 11-week intervention period.

Relevance Soldiers preparing for deployment are in need of advanced technology to help improve and optimize the functional capacity of the lumbar extensor muscles. Assuming positive results from this study and confirmatory trials, implementation of this targeted exercise protocol will maximize resilience in soldiers at high risk for low back injury, thereby helping them become more physically fit to counteract the extreme physical demands required in combat.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* Active duty soldiers in the US Army training to become combat medics at Fort Sam Houston

Exclusion Criteria:

* Cardiovascular contraindications to resistance exercise as identified by history and physical examination
* Orthopedic contraindications to resistance exercise as identified by history and physical examination
* History of systemic inflammatory disease or spinal surgery
* Low back pain intensity > "mild"
* Disability >= 50% on the Roland Morris Disability Questionnaire
* Currently receiving care for spinal pain disorder/injury
* Currently disabled due to spinal pain disorder/injury
* Currently diagnosed with or receiving treatment for a psychological or psychiatric disorder
* Currently performing progressive resistance exercises for the lumbar extensor muscles other than those included in standard for military fitness programs
* Active workers' compensation or personal injury case
* Pregnant
* Simultaneously enrolled in another biomedical clinical trial
* Drug or alcohol abuse within the past year
* Any other condition, which in the opinion of the investigators or military medical authority, would put the candidate at increased safety risk or otherwise make the candidate unsuitable for this study
* Unable or unwilling to complete the study procedures

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 582 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William S Quillen, PT,DPT,PhD, Principal Investigator — University of South Florida; John M Mayer, DC,PhD, Study Director — University of South Florida
Locations (2):
- United States (2):
  - University of South Florida, Tampa, Florida
  - Brooke Army Medical Center, Fort Sam Houston, Texas

REFERENCES:
- [Derived] Mayer JM, Childs JD, Neilson BD, Chen H, Koppenhaver SL, Quillen WS. Effect of Lumbar Progressive Resistance Exercise on Lumbar Muscular Strength and Core Muscular Endurance in Soldiers. Mil Med. 2016 Nov;181(11):e1615-e1622. doi: 10.7205/MILMED-D-15-00543. PMID 27849497

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment, enrollment, baseline assessments, and randomization procedures were completed during June 2012 through May 2013 at Fort Sam Houston, TX.
Pre-assignment Details: Assessed for eligibility: n = 698. Consented: n = 645. Deemed eligible to participate, completed baseline assessments for primary outcome, and randomized: n = 582. Reasons for ineligibility: declined to participate (n = 43), did not meet inclusion criteria (n = 28), and other or unknown reasons (n = 45).
Period: Overall Study
Arm/Group | Strengthening Exercise | Stabilization Exercise
Started | 298 | 284
Completed | 230 | 217
Not Completed | 68 | 67
Not completed — Withdrawal by Subject | 3 | 2
Not completed — academic reason | 4 | 1
Not completed — changed companies | 20 | 34
Not completed — discharged from US Army | 3 | 4
Not completed — invalid follow-up strength data | 1 | 4
Not completed — on profile | 9 | 5
Not completed — other/unknown | 28 | 17

BASELINE CHARACTERISTICS:
Population: All enrolled participants who were deemed eligible, completed baseline assessments, and were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Strengthening Exercise | Stabilization Exercise | Total
Number analyzed (Participants) | 298 | 284 | 582
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (3.8) | 21.5 (3.6) | 21.7 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 68 | 135
  Male | 231 | 216 | 447
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian | 3 | 5 | 8
  American Indian, Asian, Hispanic, White/Cau | 1 | 0 | 1
  American Indian, Black/African American, White/Cau | 1 | 0 | 1
  American Indian, White or Caucasian | 3 | 2 | 5
  Asian | 12 | 14 | 26
  Asian, Black/African American, Hispanic, White/Cau | 1 | 0 | 1
  Asian, Black or African American, Other | 1 | 0 | 1
  Asian, Hispanic | 0 | 1 | 1
  Asian, Pacific Islander | 0 | 1 | 1
  Asian, White or Caucasian | 3 | 1 | 4
  Black or African American | 27 | 26 | 53
  Black or African American, Hispanic | 1 | 0 | 1
  Black or African American, White or Caucasian | 0 | 3 | 3
  Hispanic | 46 | 41 | 87
  Hispanic, White or Caucasian | 2 | 2 | 4
  Other/unknown | 6 | 10 | 16
  Other, White or Caucasian | 1 | 0 | 1
  Pacific Islander | 2 | 4 | 6
  Pacific Islander, White or Caucasian | 0 | 2 | 2
  White or Caucasian | 188 | 172 | 360
Region of Enrollment [Number; unit: participants] — All participants were enrolled from Fort Sam Houston, TX, USA
  participants
    United States | 298 | 284 | 582
Isometric Lumbar Extension Muscular Strength [Mean (Standard Deviation); unit: Nm] — Isometric lumbar extension muscular strength (torque - Nm) as assessed by a validated physical performance test on the lumbar dynamometer
  Nm | 275.4 (87.0) | 271.7 (92.8) | 273.7 (89.9)
Isometric Core Muscular Endurance [Mean (Standard Deviation); unit: seconds] — Isometric core muscular endurance as assessed by a validated physical performance test (prone static plank test). Strengthening Exercise: n = 296; Stabilization Exercise: n = 279.
  seconds | 169.0 (62.4) | 172.8 (64.1) | 170.8 (63.2)
Dynamic Lumbar Extension Muscular Endurance [Mean (Standard Deviation); unit: repetitions] — Dynamic lumbar extension muscular endurance (# repetitions at 50% peak torque) as assessed by a validated physical performance test on the lumbar dynamometer. Strengthening Exercise: n = 285; Stabilization Exercise: n = 271.
  repetitions | 21.8 (7.7) | 22.0 (8.0) | 21.9 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Isometric Lumbar Extension Muscular Strength at 11 Weeks
Description: Isometric lumbar extension muscular strength (torque - Nm) as assessed by a validated physical performance test on the lumbar dynamometer
Time Frame: 11 weeks
Population: Adjusted (by baseline score) isometric lumbar extension muscular strength in Nm (mean ± SE) at follow-up
Measure: Mean (Standard Error); unit: Nm
Arm/Group | Strengthening Exercise | Stabilization Exercise
Number analyzed (Participants) | 230 | 217
Nm | 310.2 (6.1) | 282.7 (6.1)
Statistical Analysis 1: Comparison: Strengthening Exercise vs Stabilization Exercise; For the primary hypothesis, differences at follow-up between the two groups on lumbar extension muscular strength (Nm) were analyzed using linear mixed-effects regression models, accounting for the effects of cluster (platoon) and adjusting for baseline measures. The linear mixed-effects model treats the data as two levels (level 1 for individuals, level 2 for clusters), while also taking into account between-cluster variation; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis

2. Secondary Outcome: Isometric Core Muscular Endurance at 11 Weeks
Description: Isometric core muscular endurance as assessed by a validated physical performance test (prone static plank test)
Time Frame: 11 weeks
Population: Adjusted (by baseline score) isometric core muscular endurance in seconds (mean ± SE) at follow-up. Differences in sample sizes for this outcome (compared with primary outcome) are due to invalid test data for primary outcome (n = 4 stabilization arm; n = 1 strengthening arm), and incomplete data for this outcome (n = 1 stabilization arm).
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Strengthening Exercise | Stabilization Exercise
Number analyzed (Participants) | 231 | 220
seconds | 161.4 (7.2) | 160.2 (7.2)
Statistical Analysis 1: Comparison: Strengthening Exercise vs Stabilization Exercise; For the primary hypothesis, differences at follow-up between the two groups on core muscular endurance (seconds) were analyzed using linear mixed-effects regression models, accounting for the effects of cluster (platoon) and adjusting for baseline measures. The linear mixed-effects model treats the data as two levels (level 1 for individuals, level 2 for clusters), while also taking into account between-cluster variation; Test type: Superiority or Other; p = 0.871, Mixed Models Analysis

3. Secondary Outcome: Dynamic Lumbar Extension Muscular Endurance at 11 Weeks
Description: Dynamic lumbar extension muscular endurance (# repetitions at 50% peak torque) as assessed by a validated physical performance test on the lumbar dynamometer
Time Frame: 11 weeks
Population: Adjusted (by baseline score) isometric core muscular endurance in seconds (mean ± SE) at follow-up. Differences in sample sizes for this outcome (compared with primary outcome) are due to invalid test data for this outcome (n = 11 stabilization arm; n = 18 strengthening arm).
Measure: Mean (Standard Error); unit: repetitions
Arm/Group | Strengthening Exercise | Stabilization Exercise
Number analyzed (Participants) | 212 | 206
repetitions | 24.6 (1.0) | 21.9 (1.0)
Statistical Analysis 1: Comparison: Strengthening Exercise vs Stabilization Exercise; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event information was collected for the time frame from baseline assessments through the 11-week intervention period through the follow-up assessments, up to 12 weeks.
Arm/Group | Strengthening Exercise | Stabilization Exercise
Serious Adverse Events (participants affected / at risk) | 0/298 | 0/284
Other Adverse Events (participants affected / at risk) | 6/298 | 1/284
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strengthening Exercise (N=298) | Stabilization Exercise (N=284)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) — Low back muscle soreness following baseline lumbar extension strength test (stabilization exercise, n = 1), or following intervention session (strengthening exercise, n = 3). Mild. Related to study procedures.
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Lower extremity pain during Advanced Infantry Training and aggravated by study intervention (strengthening exercise, n = 1). Mild. Initial incident: Unrelated to study procedures. Aggravation: related to study procedures.
Musculoskeletal and connective tissue disorder - other: abdominal injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Mild. Unrelated to study procedures.
Musculoskeletal and connective tissue disorder - other: groin injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Mild. Unrelated to study procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No